CLINICAL TRIAL: NCT06091709
Title: Development, Evaluation, and Assessing the Efficacy of Multimodal Exercises and Education Tele-Rehabilitation (MEET-R) Module for Improving Pain, Posture, and Disability Level in Dentists With Work-related Low Back Pain.
Brief Title: Efficacy of Multimodal Exercises and Education Tele-Rehabilitation (MEET-R) for Low Back Pain Managment
Acronym: MEET-R
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Junaid Amin, Shahzada Junaid Amin, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEET-R for dentists with WRLBP
Record Dates: First submitted 2023-10-15; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Non-specific Low Back Pain
Keywords: Multimodal Exercises,Low back pain, Tele-Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEET-R Group (Experimental): Participants will follow the MEET-R that will include stretching, strengthening and core stabilization exercises, and education material pertaining to the proper posture during work.
  Interventions: Other: Multimodal Exercises and Education delivered through tele rehabilitation
- Control Group (Other): The control group is allowed to opt for self-care management of back pain in the form of medications, rest, conventional physiotherapy, and a home exercise plan. They are also allowed to change their self-care management during the study period; information about the use of the alternative management will be recorded. The information on self-care management will be gathered after 6 weeks at the end of the intervention
  Interventions: Other: Selafcare

INTERVENTIONS:
Other: Multimodal Exercises and Education delivered through tele rehabilitation — Participants will follow the MEET-R that will include stretching, strengthening and core stabilization exercises, and education material pertaining to the proper posture during work.
  Arms: MEET-R Group
Other: Selafcare — The control group is allowed to opt for self-care management of back pain in the form of medications, rest, conventional physiotherapy, and a home exercise plan. They are also allowed to change their self-care management during the study period; information about the use of the alternative management will be recorded. The information on self-care management will be gathered after 6 weeks at the end of the intervention
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to test the MEET-R module (Multimodal Exercises and Education Tele-Rehabilitation) for improving pain, disability, and posture of dentists with work-related non-specific chronic low back pain.

The main question is "Is MEET-R, a telerehabilitation multimodal exercises module, effective for managing pain, disability, and posture of Pakistani dentists with low back pain?" It aims to To assess the efficacy of MEET-R module for improving pain, disability, and posture of dentists with work-related non-specific chronic low back pain in a randomized controlled trial by,

1. comparing the mean difference in pain ( assessed using Numeric Rating Scale, NRS sores) before and after intervention between dentists with non-specific chronic low back pain receiving the MEET-R telerehabilitation and a control group.
2. comparing the proportion of improvement in disability, defined as having at least 30% decrease in Roland-Morris Disability Questionnaire (RMQ) score, between dentists with non-specific chronic low back pain receiving the MEET-R telerehabilitation and a control group.
3. comparing the mean difference in posture, assessed using the Rapid Entire Body Assessment (REBA) score, before and after intervention between dentists with non-specific chronic low back pain receiving the MEET-R telerehabilitation and a control group.

Intervention Group Participants will follow the MEET-R that will include stretching, strengthening and core stabilization exercises, and education material pertaining to the proper posture during work.

The Control Group The control group is allowed to opt for self-care management of back pain in the form of medications, rest, conventional physiotherapy, and a home exercise plan. They are also allowed to change their self-care management during the study period; information about the use of the alternative management will be recorded. The information on self-care management will be gathered after 6 weeks at the end of the intervention

Researchers will compare MEET-R group and control group to see if there is difference in the efficacy of MEET-R module for improving pain, disability, and posture of dentists with work-related non-specific chronic low back pain compared in a randomized controlled trial.

DETAILED DESCRIPTION:
HYPOTHESIS It is hypothesized that an innovative telerehabilitation module MEET-R that is specifically developed for dentists with work-related nonspecific chronic low back pain and approved by panelists can improve back pain, physical disability, and postural symptoms and thus, improves health-related quality of life, functioning, and satisfaction.

Research design A randomized controlled parallel group trial will be conducted to evaluate the effectiveness of MEET-R in dentists with work-related low back pain. The study protocol will adhere to the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) Study area The study participants will receive the instruction for the intervention online and be performing the intervention in their home environment under the remote supervision of a qualified physiotherapist.

Reference population

Dentist with non-specific chronic low back pain. Target population

The dentists with non-specific chronic low back pain in Lahore, Pakistan. Sampling frame

This study will include registered and practicing dentists with non-specific low back pain from private and public clinics, university clinics, and hospitals who participated in another cross-sectional study on the prevalence of MSDs in dentists in Pakistan and agreed to be contacted and participate in the trial.

Sample size calculation A sample size of 180 patients will be required for this study based on the highest sample size calculated for the primary objectives. This sample size estimation is based on the calculation of sample size in the subsequent section.

Sampling method

The participants will be selected using a simple random sampling method from a list of respondents mentioned in the sampling frame.

Randomization

Randomization will be employed to ensure that the two groups are comparable at the start of the study, and reducing the risk of selection bias. Computer-based online software (https://www.randomizer.org/) will be used to allocate the participants into intervention and control groups with a 1:2 ratio. The rationale for the ratio is described in the control group heading number 3.4.10.

Matching

In addition to randomization, matching will be used to ensure that baseline characteristics respect to the inclusion and exclusion criteria are similar between the groups. Dentists in the experimental and control groups will be matched based on variables that might affect low back pain, such as age, BMI, and severity of pain at the start of the study. Matching can help control for these variables, reducing their potential impact on the results.

Blinding The study participants will be aware of their treatment but neither intervention nor control groups will be unaware of the treatment of the other. The clinical assessment and intervention will be performed by the same investigator. That investigator will be blinded from knowing the identity of study participants by assigning codenames to the latter, derived by another investigator, and addressing them by it throughout the study. Bias and blinding are controlled by deriving different codenames for the clinical assessment and delivery of the intervention. The participants will be informed of the lack of personal address in communication during the interactive sessions. The data analyst will also be blinded to group assignments and treatment information to ensure the integrity of data analysis.

Data collection method

Step 1: (Recruitment of patients) A list of subjects identified as having low back pain including their contact information will be obtained from another (ongoing) cross-sectional study. The subjects will be approached using their contact information (WhatsApp, email, and mobile numbers) to screen their interest to participate in the trial and based on the study inclusion criteria.

Step 2 (online screening to 'confirm' diagnosis) Those meeting the first screening stage will undergo a second screening for the exclusion criteria (Irvine et al., 2015). Information on demographics, workplaces, and possible medical risk factors will also be collected.

Step 3: (Online meeting to perform physical examination) For patients who pass the second screening, an expert and registered physiotherapist will seek further a detailed history, conduct a remote physical musculoskeletal examination in an online meeting which will take 30 minutes, and assess the pain score using the NRS (Laskowski et al., 2020; Mani et al., 2017). Only patients who will meet the screening above will continue to the next step.

Step 4: (Informed consent and Baseline measurements) Each study participant will be informed about the study objective and the methods before verbal and written informed consent is sought (Figure 3). Then, the baseline assessment of the subjects will be performed to assess the primary outcomes including pain, disability levels, and posture by using the Numeric Rating Scale (NRS), Roland-Morris Disability Questionnaire, and Rapid Entire Body Assessment (REBA), respectively. In addition, the participants will be asked to complete the Patient Specific Functional Scale (PSFS) and European quality of life 5 dimensions 5 level (EQ-5D-5L) questionnaire to assess their functional status and quality of life.

Step5 (Allocation to intervention and control groups)

The subjects will be randomly assigned to the intervention and control groups (Figure 3). The intervention group will be given the link to the MEET-R which will be accessible for up to 6 weeks through a mobile application TeleHab® (VALD Health, Newstead, QLD, Australia, which is a freely available exercise prescription and tracking platform. They will be asked to follow the instruction of MEET-R throughout the 6 weeks. The MEET-R intervention included instruction on exercises, education, and ergonomics instructions in the form of an e-booklet that contains details of the instructions of their treatment protocol and a link to a video of the same information. Subsequently, reinforcement will be given periodically every week to the patients to improve their compliance and motivation by sending regular messages and telephone calls during the study period. The services provided will be free of charge throughout the study period of 6 weeks.

The control group will receive no intervention from the study and asked to continue with their existing self-care management of LBP. They will be given access to the MEET-R module after the completion of the trial.

Step 6 (Follow-up and Analysis) All the assessments made at baseline will be reassessed online after 6 weeks (Figure 3). In addition, the exercise adherence rating scale (EARS), and the Telehealth usability questionnaire (TUQ) will be assessed following the intervention. Any changes observed in the self-care management of the control group after the baseline assessment will also be recorded.

Pilot study A pilot study will also be conducted on 20 participants of the total sample to evaluate the technical, administrative, or logistic feasibility before the main trail. The justification of the pilot study is also to foresee the issues of data collection and protocol adherence. RCT will be followed by the pilot study and participants of the pilot study will be included in the RCT.

Data analysis

The data will be coded and analyzed using SPSS version 27 (PSS, Inc., Chicago, IL, USA). The categorical data will be presented in the form of frequency and percentages while continuous data will be presented as mean and standard deviation (SD). The data will be presented in the form of bar charts and pie charts. A Chi-squared test will be used to analyze associations between categorical variables. A histogram and the test of normality will be used to examine the data distribution. A paired t-test will be used for comparing pre-and post-intervention and an independent t-test for comparing intervention and control groups for normally distributed data. The significance level will be 5% for all analyses and a P-value < 0.05 will be considered a significance level.

ELIGIBILITY:
Inclusion criteria The participants must comply with the following inclusion criteria.

1) Registered and currently active practicing dentistry 2) Assessed based on history and physical examination and, diagnosed by a physiotherapist/orthopaedic/general practitioner/physiatrist to have low back pain for at least three months with pain intensity greater than 3/10 on NRC and disability level at least 5 on Roland-Morris Disability score 3) Age less than 60 years. 4) Able to read, write, and understand English 5) Have access to the internet and 6) Competent users of smartphones/laptops/tablets/pc. Exclusion criteria Additionally, the following exclusion criteria will be followed.

1. Patients who are suffering from MSDs related to other medical conditions including

   1. Neurological disorders such as spinal tumors, IVDP, spinal surgery, infection, osteoporosis, cauda equina syndrome, lumbar spine fracture, spondylolisthesis, stroke, parkinsonism and
   2. Physical disability, spinal deformities (Scoliosis, lordosis, and kyphosis), pregnancy, mental disorders, and inflammatory joint diseases (rheumatoid arthritis, gout, ankylosing spondylitis).
2. Patients who are suffering from low back pain from other causes:

   1. Back pain before practicing dentistry
   2. Has a history of trauma to the spine.
   3. Known or suspected to have serious spinal pathology.
   4. Currently undergoing a monitored exercise program or physiotherapy intervention for back pain.
   5. Any contraindication to exercise (etc. uncontrolled hypertension, respiratory and/or severe cardiac pathology)
3. Having a BMI above 35.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | From enrollment to the end of treatment at 6 weeks
  Roland-Morris Disability Questionnaire was designed to assess self-rated physical disability caused by low back pain (Jawaid et al., 2020). This validated self-report questionnaire is most sensitive for patients with mild to moderate disability due to acute, sub-acute, or chronic low back pain and assesses the physical, psychosocial, sleep and rest home management, and eating domains (Grotle, Brox, & Vollestad, 2003).
Roland-Morris Disability Questionnaire | From enrollment to the end of treatment at 6 weeks
  The Numeric Rating Scale (NRS) is the simplest and most commonly used numeric scale to measure the intensity of pain. The respondent selects a whole number and rates the pain from 0 (no pain) to 10 (worst pain). Respondents are most commonly asked to report pain intensity "in the last 24 hours". NRS is a valid and reliable scale with minimal language translation difficulties that supports the use of the NPRS across cultures and languages
Rapid Entire Body Assessment (REBA) | From enrollment to the end of treatment at 6 weeks.
  The REBA score represents the level of MSDs risk for the job task being evaluated. The minimum REBA score = 1, and the maximum REBA score = 15. As the Risk Index increases, the level of MSDs risk increases correspondingly. REBA score 1 =negligible risk, 2-3= low risk, 4-7= medium risk, 8-10= high risk, and 11 or above very high risk.

SECONDARY OUTCOMES:
Patient-Specific Functional Scale (PSFS): | From enrollment to the end of treatment at 6 weeks
  The PSFS is a self-reported and responsive outcome measure for patients with back, neck, knee, and upper extremity problems. This is a valid and reliable tool that allows patients to report on their function at baseline and follow-up. Patients are asked to rate (on an 11-point scale) the current level of difficulty associated with each activity. Following the intervention, patients are asked again to rate the activities previously identified (and are given the chance to nominate new problematic activities that might have arisen during that time)."0" represents "unable to perform" and "10" represents "able to perform at prior level"
European quality of life (EQ-5D-5L) questionnaire | From enrollment to the end of treatment at 6 weeks
  A 5-level version (EQ-5D-5L) was developed by the EuroQol Group. EQ-5D-5L is designed for self-completion by respondents, and is available in both paper and digital versions. EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
The Exercise Adherence Rating Scale (EARS) | From enrollment to the end of treatment at 6 weeks.
  The Exercise Adherence Rating Scale (EARS) is a self-reported questionnaire developed by a group of United Kingdom researchers and one of the commonly used outcome tools, which helps to identify the adherence rate of exercises and reasons for adherence and non-adherence. That is composed of six items that directly assess adherence. The six items are summed and items with positive phrases are reversely scored; meaning items 1, 4, and 6. The six items are scored using an ordinal answer scale (0 = strongly agree to 4 = disagree), with higher scores indicating greater adherence (0 to 24).
Telehealth usability questionnaire (TUQ) | From enrollment to the end of treatment at 6 weeks.
  Telehealth usability questionnaire (TUQ) consists of 21 items, evaluating treatment given through the remote rehabilitation service, software, or system.The TUQ is a comprehensive and validated tool that includes questions in the domains of usefulness, ease of use, interaction quality (effectiveness), reliability, and satisfaction. TUQ uses 7-point Likert type scale (1 = disagree and 7 = agree). The total score is calculated by summing the 21 items.

CONTACTS AND LOCATIONS:
Overall Officials: Basaruddin Ahmad, PhD, Study Director — Universiti Sains Malaysia; junaid Amin, PhD Student, Principal Investigator — Universiti Sains Malaysia